CLINICAL TRIAL: NCT00771290
Title: Prospective,Randomized Trial Comparing Colonic Distension After Intra-operative Sigmoidoscopy Using Ambient Air or Carbon Dioxide
Brief Title: Comparision of Air Versus CO2 for Distention During Sigmoidoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAB6097
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Surgery
Keywords: Rectal sparing; Colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Air insufflation with standard endoscopy unit, CO2 insufflation for colonoscopy (special CO2 insufflation unit) — comparison of Air insufflation to CO2 insufflation during intraoperative endoscopy

SUMMARY:
Intra-operative colonoscopy (inserting a flexible endoscope with a camera at its tip through the anus and up into the rectum and colon) is most often indicated to locate or verify the location of small cancer, polyp, bleeding site, or simply to inspect the bowel after the two ends have been rejoined together. Usually colonoscopy utilizes ambient air to expand and inflate the colon and, as a result, leaves the colon bloated or distended until the gas is either expelled or absorbed. This endoscopy related bowel distension is problematic in the setting of both traditional open (big incision) colorectal surgery and after minimally invasive (laparoscopic assisted) procedures.

In the case of the former, it may prove difficult to close a traditional laparotomy incision if the bowel is distended and may hinder respiration with the abdomen closed. In the setting of a laparoscopic procedure, the bowel distension limits the working space available to the surgeon. Since the laparoscopic domain is limited, a distended colon following intra-operative colonoscopy can prevent the minimally invasive completion of a case (meaning that a conversion to traditional "open" methods would be necessary) that otherwise was going well with good prospects of laparoscopic completion. Colonic distension also causes abdominal pain and lengthens the recovery time from the procedure.

The investigators believe that the use of CO2 during intra-operative colonoscopy or sigmoidoscopy (exam of only the last 2 to 2 ½ feet of the colon) will not cause long lasting bloating or distension of the colon as opposed to air. Carbon dioxide is absorbed 250 times faster than ambient air and may decrease after procedure colonic distension. This prospective, randomized study will compare the two gases in terms of colonic distension. Patients undergoing open or minimally invasive colorectal resection will be randomized to undergo intra-operative colonoscopy using one of the two gases. Direct measurements of colon diameter will be taken at specific time intervals after the colonoscopy.

DETAILED DESCRIPTION:
Colonoscopic examination of the large bowel (inserting a flexible endoscope with a camera at its tip through the anus and up into the rectum and colon) is sometimes required during a colorectal resection (abdominal operation to remove a segment or piece of colon or rectum) in order to find a small cancer, polyp, bleeding site, or simply to inspect the bowel after the two ends have been rejoined together. In order to get a good look at the large intestine with a colonoscope it is necessary to pump some gas into the colon via the scope in order to distend and inflate it. The gas that is almost universally used is room air. Since it is very hard, if not impossible, to fully suction out the gas from the colon once the exam is finished, the colon is usually quite bloated or distended after the colonoscopy. This dilatation can persist for hours or days since air is not well absorbed through the bowel wall into the body. A distended colon can cause some problems during both traditional open (big incision) surgery and laparoscopicassisted (minimally invasive) surgery. During a big incision operation, colonic distension and swelling can make it hard to close the incision at the end of the operation and can make breathing more difficult.

In contrast, during a laparoscopic procedure, the colorectal dilatation can greatly decrease the amount of working and maneuvering room that is available to the surgeon to the point where the laparoscopic approach may have to be abandoned in favor of the big incision method. Thus, colon distension following sigmoidoscopy done with air during an abdominal operation can cause problems for the patient and the surgeon.

An alternative gas that can be pumped into the colon during colonoscopy is carbon dioxide (CO2). Unlike air, CO2 is very rapidly reabsorbed into the body from the colon, about 250 times faster than air. There is now a machine available which makes it possible to easily and safely use CO2 gas to distend the colon during colonoscopy. The investigators believe that the use of CO2 during intraoperative colonoscopy or sigmoidoscopy (exam of only the last 2 to 2 ½ feet of the colon) will not cause long lasting bloating or distension of the colon as opposed to air. Patients undergoing either open (big incision) or laparoscopic (multiple small incisions) rectal or sigmoid colon resection usually need to have intraoperative sigmoidoscopy at the end of the operation to inspect the inside of the colon and rectum and to check for an air leak in the vicinity of the rejoining point (anastomosis). In this study one half of the patients will, by the flip of a coin, get CO2 during their sigmoidoscopy while the remaining half will have air used to inflated the colon during their examination. After the sigmoidoscopic exam is completed the scope will be removed, without suctioning, and the colon diameter near the rectum measured by the surgeons looking and working in the abdomen. The size of the colon will again be measured every 5 minutes for the next 20 minutes while the surgeons prepare to close the abdomen and end the surgery. At the end of the 20 minute period, if the colon remains distended, the scope will be reinserted and the excess gas suctioned out. The surgeons carrying out this study believe that the colons of those patients getting CO2 gas for the sigmoidiscopy will more rapidly shrink in size towards their original diameter than the patients who get air pumped into the colon.

ELIGIBILITY:
Inclusion Criteria:

All patients, over age 18, undergoing elective, open or minimally invasive (laparoscopicassistedor handassisted) left sided colorectal resection, for any indication, in whom it is anticipated that a transanal circular,stapled colorectal anastomosis will be constructed will be eligible for enrollment in this study, provided they are able to understand and sign the Informed Consent Form. Patients will be identified preoperatively in anticipation of undergoing the operation detailed above.

Exclusion Criteria:

Patients undergoing right sided, transverse, or descending colectomy are not eligible since their anastomosis would not be carried out with a transanally placed circular stapler. Patients undergoing abdominoperineal resection (which includes no anastomosis) are also not eligible. Patients with severe COPD or emphysema would not be eligible for entry into this study. Further, patients who are undergoing emergent surgery or elective patients who are ASA Class 3 or 4 will not be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
diameter of colon/rectal wall at surgery | at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Whelan, MD, Principal Investigator — Columbia University
Locations (1):
- NewYork Presbyterian Hospital, New York, New York, United States